CLINICAL TRIAL: NCT07222904
Title: Evaluation of the Accuracy of Patient Specific Implant in Fixation of Mandibular Sagittal Split Osteotomy
Acronym: BSSO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Principal Investigator, Eman Ashour, Assistant Lecturer at Oral and Maxillofacial Surgery department at AlAzhar University, Faculty of Dental Medicine for Girls
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OR SUR-108-2-1
Record Dates: First submitted 2025-10-27; First posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Mandible Prognathism; Mandibular Retrognathism
Keywords: Mandibular orthognathic; BSSO; Virtual planning
MeSH Terms: conditions — Malocclusion, Angle Class III

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- BSSO using PSI (Experimental): 8 Patients underwent bilateral sagittal split Osteotomy fixed with patient' specific implants
  Interventions: Device: PSI

INTERVENTIONS:
Device: PSI — orthognathic surgery BSSO using PSI

SUMMARY:
Study was Conducted on Patients were need BSSO Using PSI for reposition and fixation

DETAILED DESCRIPTION:
A prospective study was conducted, and it included 8 patients. All patients underwent mandibular sagittal split osteotomy (BSSO) using PSI for repositioning and fixation. All patients were followed up clinically for immediate,1,3,6 weeks, and 3 months postoperatively after the surgical operation to assess the occlusion, presence of numbness, bleeding, and possible temporomandibular joint (TMJ) changes. All patients underwent immediate and 3 months Ortho pantomogram, postoperative CT were superimposed to the planned preoperative CT scan to evaluate the accuracy of PSI in fixation and merging of Digital dental model to the postoperative CT scan.

ELIGIBILITY:
Inclusion Criteria:

1. Age range of patients 18-40 years old, with no gender prediction, able to read and sign the informed consent.
2. Patients with skeletal class II or class III who are in need of mandibular orthognathic surgery.

Exclusion Criteria:

1. Patients who had previous orthognathic surgery.
2. Patients with previous severe facial trauma history or fracture mandible.
3. Patients with congenital facial asymmetry.
4. Patients with systemic diseases and immunocompromised patient.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Accuracy of PSI and bony segment movements | Baseline (preoperative), immediate postoperative, and 3-month postoperative follow-up.
  Measurements using CT software after superimposition using (Mimics and 3-Matic) through fixation landmark points on both virtually planned repositioned mandible and the actual postoperative mandible, all in identical locations. Then linear measurements were performed between defined anatomical landmarks on both models using Measure distance tool, as well as between each landmark and the constructed reference planes

CONTACTS AND LOCATIONS:
Overall Officials: Hatem AlAhmady, Professor, Study Chair — Professor of maxillofacial surgery department azhar university
Locations (1):
- Eman Ashour, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No